CLINICAL TRIAL: NCT03402464
Title: Icotinib Combined With Dihydroaremisinin (DHA) Therapy in Patients With Advanced Gradually Progressed NSCLC After First-line Icotinib: an Open-label, Single-arm, Multicenter Phase II Study
Brief Title: Icotinib Combined With Dihydroaremisinin (DHA) Therapy in Patients With Advanced NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ziping Wang, professor of medicine, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV88
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: EGFR Positive Non-Small Cell Lung Cancer,Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Icotinib combined dihydroaremisinin (Experimental)
  Interventions: Drug: Icotinib combined dihydroaremisinin

INTERVENTIONS:
Drug: Icotinib combined dihydroaremisinin — Icotinib should be taken by the patients continuously until disease progressed or intolerable toxicity. On day 1-3, oral dihydroaremisinin was given at 20mg per day, the dose of dihydroaremisinin is increased to 40mg daily on day 4 to 6, and 80mg twice daily until disease progressed or intolerable toxicity.

SUMMARY:
The study was to evaluate the safety, PFS and ORR of icotinib/dihydroaremisinin (DHA)-based combination therapy in EGFR-mutated, advanced NSCLC patients who have gradually progressed disease after first-line icotinib treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients confirmed with stage IV lung adenocarcinoma by pathologic histology or cytology who can't accept surgery and radiotherapy
2. Male or female patients aged ≥18 years, life expectancy ≥ 12 weeks
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
4. Sensitive EGFR gene mutation(19/21)
5. Failed with first-line icotinib and have gradually progressed disease More than 6-month duration of first-line icotinib (from the first dosing to the imaging-confirmed progression; and discontinuation of icotinib is less than 14 days) No significantly increased tumor size compared with the final imaging evaluation

Exclusion Criteria:

1. Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease)
2. Female subjects should not be pregnant or breast-feeding
3. Patient assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol
4. Previous systemic anti-tumor therapy except for icotinib , including chemotherapy or targeted therapy ( including but not limited to monoclonal or antibodies, small molecule tyrosine kinase inhibitor, etc)
5. Tumor metastasis of the spinal cord, meninges or meningeal neoplasms confirmed by imaging or cerebrospinal fluid examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2020-09-20 (Estimated)

PRIMARY OUTCOMES:
Progress Free Survival | 18 months
Objective response rate | 18 months

SECONDARY OUTCOMES:
Overall Survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ziping Wang, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China